CLINICAL TRIAL: NCT06037421
Title: Metagenomic Analysis of Bacterial Microbiota in Breast Milk
Acronym: MIC-LAMA2
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier Sud Francilien (Other)
Responsible Party: Sponsor
Other Study IDs: 2023-A01731-44
Record Dates: First submitted 2023-09-06; First posted 2023-09-14 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Bacteria in Breast Milk
Keywords: Bacterial; newborn breast milk; neonates; infectious risk; virulence genes; agar culture methods; shotgun metagenomics; targeted metagenomics; microbiota
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Human breast milk samples, mother's stool samples, infant's stool samples, mother's saliva samples, infant's saliva samples, mother's skin samples, mother's blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Human breast milk sampling — Human breast milk sampling
Other: Saddle sampling — Saddle sampling
Other: Skin sampling — Skin sampling
Other: Saliva sampling — Saliva sampling
Other: blood sampling — blood sampling

SUMMARY:
The aim of this study is to determine the extent to which bacteria in the breast milk microbiota represent an infectious risk for premature infants, by investigating whether they possess virulence genes, and if so, whether these are expressed or repressed.

DETAILED DESCRIPTION:
There are still many unknowns about the exact bacterial composition of breast milk, and the theoretical and real risks represented by its microbiota. In addition to determining the Total Aerobic Flora (TAF) and the Staphylococcus aureus presence, the most commonly isolated enterobacterales species identified by agar culture by the Prevention and Infection Control department are also among those potentially found in diagnostic samples: Enterobacter cloacae, Klebsiella pneumoniae, Klebsiella aerogenes, Klebsiella oxytoca and Escherichia coli. However, it is not yet known whether these are identical strains or not. It is therefore legitimate to ask whether there are any differences between the strains present in the microbiota of breast milk and those responsible for newborn infections.

Conventional methods for enumerating and identifying the bacteria making up the milk microbiota are not standardized, which makes it difficult to draw up a precise, multicentric inventory of its composition. It is therefore impossible to know whether exceeding a threshold value defined by expert consensus represents a real danger for newborns who must receive breast milk.

At the Centre National de Recherche en Génomique Humaine (CNRGH), a metagenomic sequencing approach makes it possible to study the microbiota using two complementary methodologies. Either by sequencing the genomes of organisms (bacteria, viruses, fungi, etc.) present in the environment to be analyzed (shotgun metagenomics), or by sequencing one or more genes specific to each bacterial species (targeted metagenomics). The gene that codes for 16S ribosomal RNA (rRNA) has sequence regions common to different bacterial species, as well as variable regions that can be used to distinguish the bacteria present in a sample.

A comparison of the composition of the bacterial microbiota in breast milk using conventional agar culture methods and metagenomic analysis methods would enable us to make progress in understanding its potential involvement in infectious pathologies in premature infants. It is in this scientific and medical context that a collaborative project was initiated for the first time between the departments of Neonatal Medicine and Intensive Care and of Prevention and Infection Control, and the CNRGH. This was a pilot study with the aim of perpetuating this collaboration, which combines scientific knowledge of the metagenome with the CNRGH's high-performance technological tools, as well as potential applications in the medical environment in the CHSF's care departments.

ELIGIBILITY:
Inclusion Criteria:

* Women of legal age who have given birth at the CHSF (or in another establishment) and whose newborn(s) are being cared for in the CHSF's Neonatal Medicine and Intensive Care Unit,
* Women wishing to give their milk to their child,
* Parents who have given their consent for the mother-child couple to take part in the study.

Exclusion Criteria:

* Mother having received antibiotic therapy in the 3 months prior to delivery, except for those who received injectable antibiotic prophylaxis during delivery.

Min Age: 1 Hour | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Mother-infant pairs whose newborn(s) are being cared for in the CHSF's Neonatal Medicine and Intensive Care Unit.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2025-09-08 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Assessing the potential pathogenic risk of certain bacteria in breast milk. | at day 0
  Presence of virulence genes in strains of bacteria with pathogenic potential (S. aureus, K. aerogenes, E. coli, K. pneumoniae, K. oxytoca, E. cloacae) in breast milk.

OTHER OUTCOMES:
Comparing the microbial ecologies of breast milk by bacterial culture and metagenomics. | at day 0
  Presence in breast milk of identical bacterial genera or species/strains between sequencing and bacterial culture.
If bacteria isolated from breast milk contain virulence genes, establish whether they are activated or repressed. | at day 0
  Production by bacteria isolated from breast milk of the mRNA and/or protein corresponding to the virulence gene(s) identified.
Establish whether strains of bacteria with pathogenic potential (S. aureus, K. aerogenes, E. coli, K. pneumoniae, K. oxytoca, E. cloacae) found in breast milk contain antibiotic resistance genes. | at day 0
  Presence of antibiotic resistance genes in strains of bacteria with pathogenic potential (S. aureus, K. aerogenes, E. coli, K. pneumoniae, K. oxytoca, E. cloacae) found in breast milk.
If so, establish whether these are activated or repressed. | at day 0
  Production by bacteria isolated from breast milk of the mRNA and/or protein corresponding to the antibiotic resistance gene.
Compare the microbial ecology of different ecosystems: intestinal, oral and cutaneous with that of breast milk, using bacterial culture and metagenomics. | at day 0
  Presence of common bacteria in different samples (child's stool and saliva + mother's stool, saliva, skin swab and milk).
Check maternal blood for the presence of essentially anaerobic bacteria such as bifidobacteria and/or mononuclear cells such as dendritic cells or macrophages, a potential reflection of the entero-mammary pathway. | at day 0
  Presence of mainly anaerobic bifidobacteria and/or mononuclear dendritic cells in maternal blood; biological marker of the entero-mammary tract.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Sud Francilien, Corbeil-Essonnes, France, France

IPD SHARING:
Plan to Share IPD: No